CLINICAL TRIAL: NCT03414723
Title: An Open Label, 2-treatment, 2-period, Single Sequence Study to Evaluate Pharmacokinetic Drug-drug Interaction Between Ramipril and Sotagliflozin at Steady State in Healthy Subjects
Brief Title: A Drug-Drug Interaction Study Between Sotagliflozin and Ramipril
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: INT14935; 2017-002650-37; U1111-1196-5355 (Other: UTN)
Record Dates: First submitted 2018-01-18; First posted 2018-01-30 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus; Healthy Subjects
MeSH Terms: conditions — Diabetes Mellitus | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SAR439954 with or without ramipril (Experimental): * On Period 1, following an overnight fast, subjects will receive once daily single morning oral intake of sotagliflozin from Day 1 to Day 5 followed by the first meal that has to be started within 10 min after dosing.
  * On Day 1 of the Period 2, study subjects will begin a 10-day ramipril regimen following an overnight fast. From Day 6 to Day 10, subjects will receive once daily single morning oral intake of ramipril concomitantly to the sotagliflozin dosing.
  Interventions: Drug: Sotagliflozin (SAR439954); Drug: Ramipril

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: tablets
  Route of administration: oral
Drug: Ramipril — Pharmaceutical form: tablets
  Route of administration: oral

SUMMARY:
Primary Objective:

To evaluate the effects of multiple-dose ramipril on the steady state pharmacokinetic (PK) parameters of sotagliflozin and its main metabolite (sotagliflozin-3-O-glucuronide) in healthy male and female subjects.

Secondary Objectives:

* To assess the effects of multiple-dose sotagliflozin on the PK of ramipril and its active metabolite (ramiprilat).
* To assess the safety and tolerability of multiple-dose sotagliflozin with and without multiple-dose of ramipril.

DETAILED DESCRIPTION:
The expected duration of subject participation, including Screening of up to 29 days, Treatment Periods of 6 days and 11 days each with a Washout period of minimum of 7 days in between periods, Follow-up period of 6 days, and end-of-study-period of 10-14 days after last sotagliflozin dose, is approximately 66 days.

ELIGIBILITY:
Inclusion criteria :

* Healthy male or female subjects, between 18 and 55 years of age, inclusive.
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index between 18.0 and 32.0 kg/m², inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs after 10 minutes resting in supine position:
* 100 mmHg <systolic blood pressure (SBP) <140 mmHg,
* 60 mmHg <diastolic blood pressure (DBP) <90 mmHg,
* 50 bpm <heart rate (HR) <90 bpm.
* Standard 12-lead electrocardiogram (ECG) parameters after 10 minutes resting in supine position in the following ranges; 120 ms<PR<200 ms, QRS <120 ms, QTc ≤430 ms if male and QTc ≤450 ms if female with normal ECG tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant.
* Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy subjects; however serum creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase) should be strictly below the ULN. Total bilirubin out of normal range can be acceptable if total bilirubin should not exceed 1.5 the upper limit with normal conjugated bilirubin values (unless the subject has documented Gilbert syndrome).
* Female subject must use a double contraception method including a highly effective method of birth control except if she has undergone sterilization at least 3 months earlier or is postmenopausal. The accepted double contraception methods include the use of 1 of the following contraceptive options: (1) intrauterine device; (2) condom or diaphragm or cervical/vault cap, in addition to spermicide. Menopause is defined as being amenorrheic for at least 2 years with plasma follicle stimulating hormone (FSH) value being within the normal range for postmenopausal women according to the local laboratory. Hormonal contraception is NOT acceptable in this study due to drug interaction.
* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* History of renal disease, or significant abnormal kidney function test with glomerular filtration rate (GFR) <90 mL/min as calculated using the Cockcroft-Gault equation.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation, any volume, within 2 months before inclusion.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis).
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day)
* If female, pregnancy (defined as positive β-HCG blood test if applicable), breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion. Any oral contraceptives during the screening period or for at least 15 days prior to inclusion; any injectable contraceptives or hormonal intrauterine devices within 12 months prior to inclusion; or topical controlled delivery contraceptives (patch) for 3 months prior to inclusion.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
Assessment of PK parameter: AUCtau | On Day 10 (Period 2)
  Sotagliflozin with ramipril: Area under the curve (AUC) to the end of the dosing period (AUCtau)
Assessment of PK parameter: AUCtau | On Day 5 (Period 1)
  Sotagliflozin without ramipril: AUCtau

SECONDARY OUTCOMES:
Assessment of PK parameter: Cmax | On Day 10 (Period 2)
  Sotagliflozin with ramipril: Maximum plasma concentration (Cmax)
Assessment of PK parameter: Cmax | On Day 5 (Period 1)
  Sotagliflozin without ramipril: Cmax
Assessment of PK parameter: tmax | On Day 10 (Period 2)
  Sotagliflozin with ramipril: Time to reach Cmax (tmax)
Assessment of PK parameter: tmax | On Day 5 (Period 1)
  Sotagliflozin without ramipril: tmax
Adverse events | Up to Day 37
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 2760001, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org